CLINICAL TRIAL: NCT00092521
Title: A Study to Evaluate the Efficacy of Quadrivalent HPV Vaccine in Reducing the Incidence of HPV 6-, 11-, 16-, and 18-Related CIN, AIS, and Cervical Cancer, and HPV 6-, 11-, 16-, and 18-Related External Genital Warts, Vulvar Intraepithelial Neoplasia Vaginal Intraepithelial Neoplasia, Vulvar Cancer, and Vaginal Cancer in 16- to 23-Year-Old Women
Brief Title: Cervical Intraepithelial Neoplasm (CIN)-Warts Efficacy Trial in Women (Gardasil)(V501-013)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-013; 2004_081
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Results first posted 2009-11-20 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Cervical Cancer; Genital Warts
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): V501
  Interventions: Biological: V501
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: Placebo
- 3 (Experimental): HPV 16 Monovalent Vaccine
  Interventions: Biological: Human Papillomavirus (HPV) 16 Monovalent

INTERVENTIONS:
Biological: V501 — Final Manufactured Product (FMP) quadrivalent HPV vaccine, a 0.5 mL intramuscular injection given at Day 1, Month 2 and Month 6.
  Arms: 1
Biological: Comparator: Placebo — a 0.5 mL intramuscular placebo injection given at Day 1, Month 2 and Month 6.
  Arms: 2
Biological: Human Papillomavirus (HPV) 16 Monovalent — HPV 16 Monovalent vaccine, a 0.5 mL intramuscular injection given at Day 1, Month 2 and Month 6.
  Arms: 3

SUMMARY:
The primary purpose of the study is to determine if GARDASIL (V501) with four components is able to prevent cervical cancer, cervical dysplasia, including Cervical Intraepithelial Neoplasia (CIN)(Any Grade) and Adenocarcinoma In Situ (AIS), and genital warts.

ELIGIBILITY:
Inclusion Criteria:

* Female with an intact uterus with lifetime history of 0-4 sexual partners

Exclusion Criteria:

* Prior Human Papillomavirus (HPV) vaccination
* Prior abnormal paps
* History of genital warts

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5759 (Actual)
Dates: Start 2001-12; Primary Completion 2007-07 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Garland SM, Steben M, Sings HL, James M, Lu S, Railkar R, Barr E, Haupt RM, Joura EA. Natural history of genital warts: analysis of the placebo arm of 2 randomized phase III trials of a quadrivalent human papillomavirus (types 6, 11, 16, and 18) vaccine. J Infect Dis. 2009 Mar 15;199(6):805-14. doi: 10.1086/597071. PMID 19199546
- [Background] Barr E, Gause CK, Bautista OM, Railkar RA, Lupinacci LC, Insinga RP, Sings HL, Haupt RM. Impact of a prophylactic quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like particle vaccine in a sexually active population of North American women. Am J Obstet Gynecol. 2008 Mar;198(3):261.e1-11. doi: 10.1016/j.ajog.2007.09.001. PMID 18313445
- [Background] Garland SM, Hernandez-Avila M, Wheeler CM, Perez G, Harper DM, Leodolter S, Tang GW, Ferris DG, Steben M, Bryan J, Taddeo FJ, Railkar R, Esser MT, Sings HL, Nelson M, Boslego J, Sattler C, Barr E, Koutsky LA; Females United to Unilaterally Reduce Endo/Ectocervical Disease (FUTURE) I Investigators. Quadrivalent vaccine against human papillomavirus to prevent anogenital diseases. N Engl J Med. 2007 May 10;356(19):1928-43. doi: 10.1056/NEJMoa061760. PMID 17494926
- [Background] Joura EA, Leodolter S, Hernandez-Avila M, Wheeler CM, Perez G, Koutsky LA, Garland SM, Harper DM, Tang GW, Ferris DG, Steben M, Jones RW, Bryan J, Taddeo FJ, Bautista OM, Esser MT, Sings HL, Nelson M, Boslego JW, Sattler C, Barr E, Paavonen J. Efficacy of a quadrivalent prophylactic human papillomavirus (types 6, 11, 16, and 18) L1 virus-like-particle vaccine against high-grade vulval and vaginal lesions: a combined analysis of three randomised clinical trials. Lancet. 2007 May 19;369(9574):1693-702. doi: 10.1016/S0140-6736(07)60777-6. PMID 17512854
- [Background] Insinga RP, Dasbach EJ, Allen SE, Carides GW, Myers ER. Reductions in human papillomavirus-disease resource use and costs with quadrivalent human papillomavirus (types 6, 11, 16, and 18) recombinant vaccination: the FUTURE Study Economic Evaluation. Value Health. 2008 Dec;11(7):1022-32. doi: 10.1111/j.1524-4733.2008.00342.x. Epub 2008 May 16. PMID 18489503
- [Background] Perez G, Lazcano-Ponce E, Hernandez-Avila M, Garcia PJ, Munoz N, Villa LL, Bryan J, Taddeo FJ, Lu S, Esser MT, Vuocolo S, Sattler C, Barr E. Safety, immunogenicity, and efficacy of quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like-particle vaccine in Latin American women. Int J Cancer. 2008 Mar 15;122(6):1311-8. doi: 10.1002/ijc.23260. PMID 18000825
- [Background] FUTURE II Study Group. Prophylactic efficacy of a quadrivalent human papillomavirus (HPV) vaccine in women with virological evidence of HPV infection. J Infect Dis. 2007 Nov 15;196(10):1438-46. doi: 10.1086/522864. Epub 2007 Oct 31. PMID 18008221
- [Background] Ault KA; Future II Study Group. Effect of prophylactic human papillomavirus L1 virus-like-particle vaccine on risk of cervical intraepithelial neoplasia grade 2, grade 3, and adenocarcinoma in situ: a combined analysis of four randomised clinical trials. Lancet. 2007 Jun 2;369(9576):1861-1868. doi: 10.1016/S0140-6736(07)60852-6. PMID 17544766
- [Background] Giuliano AR, Lazcano-Ponce E, Villa L, Nolan T, Marchant C, Radley D, Golm G, McCarroll K, Yu J, Esser MT, Vuocolo SC, Barr E. Impact of baseline covariates on the immunogenicity of a quadrivalent (types 6, 11, 16, and 18) human papillomavirus virus-like-particle vaccine. J Infect Dis. 2007 Oct 15;196(8):1153-62. doi: 10.1086/521679. Epub 2007 Sep 17. PMID 17955433
- [Background] Garland SM, Insinga RP, Sings HL, Haupt RM, Joura EA. Human papillomavirus infections and vulvar disease development. Cancer Epidemiol Biomarkers Prev. 2009 Jun;18(6):1777-84. doi: 10.1158/1055-9965.EPI-09-0067. PMID 19505910
- [Derived] Joura E, Kjaer SK, Bautista O, Luxembourg A, Saah A, Giuliano A. Effect of Prior 9-Valent Human Papillomavirus Vaccination on Subsequent Lower Genital Tract Dysplasia After Cervical Excisional Surgery. Obstet Gynecol. 2026 Jan 1;147(1):73-82. doi: 10.1097/AOG.0000000000006113. Epub 2025 Oct 30. PMID 41166720
- [Derived] Doshi P, Bourgeois F, Hong K, Jones M, Lee H, Shamseer L, Spence O, Jefferson T. Adjuvant-containing control arms in pivotal quadrivalent human papillomavirus vaccine trials: restoration of previously unpublished methodology. BMJ Evid Based Med. 2020 Dec;25(6):213-219. doi: 10.1136/bmjebm-2019-111331. Epub 2020 Mar 17. PMID 32184277
- [Derived] Giuliano AR, Joura EA, Garland SM, Huh WK, Iversen OE, Kjaer SK, Ferenczy A, Kurman RJ, Ronnett BM, Stoler MH, Bautista OM, Moeller E, Ritter M, Shields C, Luxembourg A. Nine-valent HPV vaccine efficacy against related diseases and definitive therapy: comparison with historic placebo population. Gynecol Oncol. 2019 Jul;154(1):110-117. doi: 10.1016/j.ygyno.2019.03.253. Epub 2019 Apr 11. PMID 30982556
- [Derived] Garland SM, Joura EA, Ault KA, Bosch FX, Brown DR, Castellsague X, Ferenczy A, Ferris DG, Giuliano AR, Hernandez-Avila M, Huh WK, Iversen OE, Kjaer SK, Kurman RJ, Luna J, Monsonego J, Munoz N, Paavonen J, Pitisuttihum P, Ronnett BM, Steben M, Stoler MH, Wheeler CM, Wiley DJ, Perez G, Saah AJ, Luxembourg A, Li S, DiNubile MJ, Wagner M, Velicer C. Human Papillomavirus Genotypes From Vaginal and Vulvar Intraepithelial Neoplasia in Females 15-26 Years of Age. Obstet Gynecol. 2018 Aug;132(2):261-270. doi: 10.1097/AOG.0000000000002736. PMID 29995724
- [Derived] Castellsague X, Ault KA, Bosch FX, Brown D, Cuzick J, Ferris DG, Joura EA, Garland SM, Giuliano AR, Hernandez-Avila M, Huh W, Iversen OE, Kjaer SK, Luna J, Monsonego J, Munoz N, Myers E, Paavonen J, Pitisuttihum P, Steben M, Wheeler CM, Perez G, Saah A, Luxembourg A, Sings HL, Velicer C. Human papillomavirus detection in cervical neoplasia attributed to 12 high-risk human papillomavirus genotypes by region. Papillomavirus Res. 2016 Dec;2:61-69. doi: 10.1016/j.pvr.2016.03.002. Epub 2016 Mar 14. PMID 29074187
- [Derived] Clark LR, Myers ER, Huh W, Joura EA, Paavonen J, Perez G, James MK, Sings HL, Haupt RM, Saah AJ, Garner EI. Clinical trial experience with prophylactic human papillomavirus 6/11/16/18 vaccine in young black women. J Adolesc Health. 2013 Mar;52(3):322-9. doi: 10.1016/j.jadohealth.2012.07.003. Epub 2012 Aug 15. PMID 23299013
- [Derived] Ruiz AM, Ruiz JE, Gavilanes AV, Eriksson T, Lehtinen M, Perez G, Sings HL, James MK, Haupt RM; FUTURE I and II Study Group. Proximity of first sexual intercourse to menarche and risk of high-grade cervical disease. J Infect Dis. 2012 Dec 15;206(12):1887-96. doi: 10.1093/infdis/jis612. Epub 2012 Oct 12. PMID 23066159
- [Derived] Joura EA, Garland SM, Paavonen J, Ferris DG, Perez G, Ault KA, Huh WK, Sings HL, James MK, Haupt RM; FUTURE I and II Study Group. Effect of the human papillomavirus (HPV) quadrivalent vaccine in a subgroup of women with cervical and vulvar disease: retrospective pooled analysis of trial data. BMJ. 2012 Mar 27;344:e1401. doi: 10.1136/bmj.e1401. PMID 22454089
- [Derived] Haupt RM, Wheeler CM, Brown DR, Garland SM, Ferris DG, Paavonen JA, Lehtinen MO, Steben M, Joura EA, Giacoletti KE, Radley DR, James MK, Saah AJ, Sings HL; FUTURE I and II Investigators. Impact of an HPV6/11/16/18 L1 virus-like particle vaccine on progression to cervical intraepithelial neoplasia in seropositive women with HPV16/18 infection. Int J Cancer. 2011 Dec 1;129(11):2632-42. doi: 10.1002/ijc.25940. Epub 2011 Apr 13. PMID 21491420
- [Derived] Lehtinen M, Ault KA, Lyytikainen E, Dillner J, Garland SM, Ferris DG, Koutsky LA, Sings HL, Lu S, Haupt RM, Paavonen J; FUTURE I and II Study Group. Chlamydia trachomatis infection and risk of cervical intraepithelial neoplasia. Sex Transm Infect. 2011 Aug;87(5):372-6. doi: 10.1136/sti.2010.044354. Epub 2011 Apr 6. PMID 21471141
- [Derived] Ault KA, Joura EA, Kjaer SK, Iversen OE, Wheeler CM, Perez G, Brown DR, Koutsky LA, Garland SM, Olsson SE, Tang GW, Ferris DG, Paavonen J, Steben M, Bosch FX, Majewski S, Munoz N, Sings HL, Harkins K, Rutkowski MA, Haupt RM, Garner EI; FUTURE I and II Study Group. Adenocarcinoma in situ and associated human papillomavirus type distribution observed in two clinical trials of a quadrivalent human papillomavirus vaccine. Int J Cancer. 2011 Mar 15;128(6):1344-53. doi: 10.1002/ijc.25723. Epub 2011 Jan 12. PMID 20949623
- [Derived] FUTURE I/II Study Group; Dillner J, Kjaer SK, Wheeler CM, Sigurdsson K, Iversen OE, Hernandez-Avila M, Perez G, Brown DR, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Lehtinen M, Steben M, Bosch FX, Joura EA, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan JT, Maansson R, Lu S, Vuocolo S, Hesley TM, Barr E, Haupt R. Four year efficacy of prophylactic human papillomavirus quadrivalent vaccine against low grade cervical, vulvar, and vaginal intraepithelial neoplasia and anogenital warts: randomised controlled trial. BMJ. 2010 Jul 20;341:c3493. doi: 10.1136/bmj.c3493. PMID 20647284
- [Derived] Garland SM, Ault KA, Gall SA, Paavonen J, Sings HL, Ciprero KL, Saah A, Marino D, Ryan D, Radley D, Zhou H, Haupt RM, Garner EIO; Quadrivalent Human Papillomavirus Vaccine Phase III Investigators. Pregnancy and infant outcomes in the clinical trials of a human papillomavirus type 6/11/16/18 vaccine: a combined analysis of five randomized controlled trials. Obstet Gynecol. 2009 Dec;114(6):1179-1188. doi: 10.1097/AOG.0b013e3181c2ca21. PMID 19935017
- [Derived] Brown DR, Kjaer SK, Sigurdsson K, Iversen OE, Hernandez-Avila M, Wheeler CM, Perez G, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Steben M, Bosch FX, Dillner J, Joura EA, Kurman RJ, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan J, Lupinacci LC, Giacoletti KE, Sings HL, James M, Hesley TM, Barr E. The impact of quadrivalent human papillomavirus (HPV; types 6, 11, 16, and 18) L1 virus-like particle vaccine on infection and disease due to oncogenic nonvaccine HPV types in generally HPV-naive women aged 16-26 years. J Infect Dis. 2009 Apr 1;199(7):926-35. doi: 10.1086/597307. PMID 19236279
- [Derived] Wheeler CM, Kjaer SK, Sigurdsson K, Iversen OE, Hernandez-Avila M, Perez G, Brown DR, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Steben M, Bosch FX, Dillner J, Joura EA, Kurman RJ, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan J, Lupinacci LC, Giacoletti KE, James M, Vuocolo S, Hesley TM, Barr E. The impact of quadrivalent human papillomavirus (HPV; types 6, 11, 16, and 18) L1 virus-like particle vaccine on infection and disease due to oncogenic nonvaccine HPV types in sexually active women aged 16-26 years. J Infect Dis. 2009 Apr 1;199(7):936-44. doi: 10.1086/597309. PMID 19236277
- [Derived] Six L, Leodolter S, Sings HL, Barr E, Haupt R, Joura EA. Prevalence of human papillomavirus types 6, 11, 16 and 18 in young Austrian women - baseline data of a phase III vaccine trial. Wien Klin Wochenschr. 2008;120(21-22):666-71. doi: 10.1007/s00508-008-1093-3. PMID 19116707
- [Derived] Wheeler CM, Bautista OM, Tomassini JE, Nelson M, Sattler CA, Barr E; Protocol 11 study Investigators. Safety and immunogenicity of co-administered quadrivalent human papillomavirus (HPV)-6/11/16/18 L1 virus-like particle (VLP) and hepatitis B (HBV) vaccines. Vaccine. 2008 Jan 30;26(5):686-96. doi: 10.1016/j.vaccine.2007.11.043. Epub 2007 Dec 5. PMID 18164106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study Protocol 013 (NCT00092521) (N =5759 total randomized) was comprised of two sub-studies: Protocol 011 (NCT00517309) (N=1877 total randomized) and Protocol 012 (NCT00092482) (N=3882 total randomized). Final safety data are presented in the results for Protocol 013 (NCT00092521): the final participant visit took place on 19 January 2009.
Groups:
- Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine: The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 1 were vaccinated (at Day 1, Month 2 and Month 6) with the Quadrivalent Human papillomavirus (HPV) vaccine.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the Quadrivalent HPV vaccine; from completion of the Vaccination Period at Month 7 through Month 48 of the study.
- Group 2 - Base Study Monovalent HPV (Type 16) Vaccine: The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 2 were vaccinated (at Day 1, Month 2 and Month 6) with the Monovalent (HPV 16) HPV vaccine.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the Monovalent (HPV 16) HPV vaccine; from completion of the Vaccination Period at Month 7 through Month 48 of the study.
  Group 2 Base Study Monovalent HPV (Type 16) Vaccine was not part of the pre-specified efficacy analysis population.
- Group 3 - Base Study Placebo: The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 3 were vaccinated (at Day 1, Month 2 and Month 6) with placebo.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received placebo; from completion of the Vaccination Period at Month 7 through Month 48 of the study.
- Group 4 - Quadrivalent Human Papillomavirus Vaccine Extension: This group includes subjects who entered the extension including subjects who in the base study received fewer than the full three doses of Quadrivalent HPV vaccine during the base study (i.e., subjects who received placebo in the base study; subjects who received monovalent [type 16] HPV vaccine in the base study, or subjects who received <=2 doses of quadrivalent HPV vaccine in the base study). Subjects who discontinued the base portion of the study could enter the extension portion of the study. In the extension period subjects designated as "Completed Period" are those who received three doses of quadrivalent HPV vaccine and completed all required follow-up visits. Subjects designated as "Not Completed" are those who: a) Received all three vaccinations, but did not complete follow-up; b) Did not receive all vaccinations, but completed follow-up, or c) Did not receive all vaccinations, and did not complete follow-up.
Period: Vaccination (Day 1 Through Month 7)
Arm/Group | Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine | Group 2 - Base Study Monovalent HPV (Type 16) Vaccine | Group 3 - Base Study Placebo | Group 4 - Quadrivalent Human Papillomavirus Vaccine Extension
Started | 2723 | 304 | 2732 | 0
Completed | 2583 | 290 | 2586 | 0
Not Completed | 140 | 14 | 146 | 0
Not completed — Randomized Not Vaccinated | 6 | 0 | 7 | 0
Not completed — Adverse Event | 1 | 0 | 7 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 51 | 6 | 44 | 0
Not completed — Pregnancy | 5 | 0 | 7 | 0
Not completed — Withdrawal by Subject | 59 | 7 | 62 | 0
Not completed — Moved | 14 | 1 | 18 | 0
Not completed — Unblinded | 2 | 0 | 0 | 0
Not completed — New Medical History (Not AE) | 2 | 0 | 0 | 0
Period: Follow-Up (After Month 7)
Arm/Group | Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine | Group 2 - Base Study Monovalent HPV (Type 16) Vaccine | Group 3 - Base Study Placebo | Group 4 - Quadrivalent Human Papillomavirus Vaccine Extension
Started | 2599 (Includes subjects who did not receive 3 doses of vaccine/placebo but continued into the follow-up) | 291 (Includes subjects who did not receive 3 doses of vaccine/placebo but continued into the follow-up) | 2607 (Includes subjects who did not receive 3 doses of vaccine/placebo but continued into the follow-up) | 0
Completed | 2353 | 155 | 1959 | 0
Not Completed | 246 | 136 | 648 | 0
Not completed — Subjects Continuing | 34 | 4 | 35 | 0
Not completed — Subjects in Extension | 13 | 109 | 412 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 113 | 14 | 108 | 0
Not completed — Protocol Violation | 1 | 1 | 5 | 0
Not completed — Withdrawal by Subject | 40 | 6 | 51 | 0
Not completed — Moved | 32 | 2 | 28 | 0
Not completed — Site Terminated | 3 | 0 | 3 | 0
Not completed — Travel | 2 | 0 | 0 | 0
Not completed — Visits Compressed | 5 | 0 | 5 | 0
Period: Extension Study (Group 4)
Arm/Group | Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine | Group 2 - Base Study Monovalent HPV (Type 16) Vaccine | Group 3 - Base Study Placebo | Group 4 - Quadrivalent Human Papillomavirus Vaccine Extension
Started | 0 | 0 | 0 | 844
Initiated Extension Study | 0 | 0 | 0 | 829
Received >=1 Dose in Extension Study | 0 | 0 | 0 | 801
Completed | 0 | 0 | 0 | 635
Not Completed | 0 | 0 | 0 | 209
Not completed — Excluded ineligible for extension | 0 | 0 | 0 | 23
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 87
Not completed — Pregnancy | 0 | 0 | 0 | 4
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 46
Not completed — Moved | 0 | 0 | 0 | 16
Not completed — Site Terminated | 0 | 0 | 0 | 4
Not completed — Unable/unwilling to return | 0 | 0 | 0 | 25

BASELINE CHARACTERISTICS:
Groups:
- Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine: The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 1 were vaccinated (at Day 1, Month 2 and Month 6) with the Quadrivalent HPV vaccine.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the Quadrivalent HPV vaccine; from completion of the Vaccination Period at Month 7 through Month 48 of the study.
- Group 2 - Base Study Monovalent HPV (Type 16) Vaccine: The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 2 were vaccinated (at Day 1, Month 2 and Month 6) with the Monovalent (HPV 16) HPV vaccine.
  The Follow-up Period for the Base Study encompassed the follow-up of subjects who had received the Monovalent (HPV 16) HPV vaccine; from completion of the Vaccination Period at Month 7 through Month 48 of the study.
- Total: Total of all reporting groups
Arm/Group | Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine | Group 2 - Base Study Monovalent HPV (Type 16) Vaccine | Group 3 - Base Study Placebo | Total
Number analyzed (Participants) | 2723 | 304 | 2732 | 5759
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.2 (1.8) | 20.2 (1.74) | 20.3 (1.8) | 20.3 (1.8)
Age, Continuous [Median (Full Range); unit: Years] | 20 [16 to 24] | 20 [16 to 24] | 20 [16 to 24] | 20 [16 to 24]
Age, Customized [Number; unit: Participants] — Although the upper age limit for this study was 23 years old, four subjects aged 24 were randomized into the study.
  Participants
    16 to 24 Years of Age | 2723 | 304 | 2732 | 5759
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2723 | 304 | 2732 | 5759
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 151 | 27 | 165 | 343
  Black | 136 | 5 | 167 | 308
  Hispanic American | 567 | 93 | 566 | 1226
  Native American | 10 | 2 | 10 | 22
  White | 1600 | 171 | 1558 | 3329
  Other - Unspecified | 259 | 6 | 266 | 531

OUTCOME MEASURES:

1. Primary Outcome: Incidence of HPV 6/11/16/18-related Cervical Intraepithelial Neoplasia (CIN)(Any Grade), Adenocarcinoma In Situ (AIS) or Cervical Cancer
Time Frame: Follow-up through end of study (4 years)
Population: Per-protocol population: subjects must have no major protocol violations, must be seronegative to the relevant type at Day 1 and Polymerase Chain Reaction (PCR) negative to the relevant type through Month 7, and must provide follow-up data. Group 2 Base Study Monovalent HPV Vaccine was not part of the pre-specified efficacy analysis population.
Measure: Number; unit: incidence rate per 100 person-years
Arm/Group | Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine | Group 3 - Base Study Placebo
Number analyzed (Participants) | 2241 | 2258
incidence rate per 100 person-years | 0 | 1.2
Statistical Analysis 1: Comparison: Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine vs Group 3 - Base Study Placebo; Test type: Superiority or Other; Percent relative risk reduction = 100, 95% CI [95.1 to 100] — Confidence Interval (CI) based on binomial tail probabilities and not from a dispersion parameter

2. Primary Outcome: Incidence of HPV 6/11/16/18-related External Genital Lesions (EGL) [Genital Warts, Vulvar/Vaginal Intraepithelial Neoplasia (Any Grade), Vulvar/Vaginal Cancer]
Time Frame: Follow-up through end of study (4 years)
Population: Per-protocol population: subjects must have no major protocol violations, must be seronegative to the relevant type at Day 1 and PCR negative to the relevant type through Month 7, and must provide follow-up data.
  Group 2 Base Study Monovalent HPV (Type 16) Vaccine was not part of the pre-specified efficacy analysis population.
Measure: Number; unit: incidence rate per 100 person-years
Arm/Group | Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine | Group 3 - Base Study Placebo
Number analyzed (Participants) | 2261 | 2279
incidence rate per 100 person-years | 0 | 1.1
Statistical Analysis 1: Comparison: Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine vs Group 3 - Base Study Placebo; Test type: Superiority or Other; Percent relative risk reduction = 100, 95% CI [94.9 to 100] — CI based on binomial tail probabilities and not from a dispersion parameter

ADVERSE EVENTS:
Description: Number of subjects at risk included randomized subjects who had follow-up. For Group 4 (Extension), number of subjects at risk included those who received >=1 vaccination in the extension study. Both serious and Other AEs were collected in the base period and only serious AEs were collected in the extension period.
Arm/Group | Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine | Group 2 - Base Study Monovalent HPV (Type 16) Vaccine | Group 3 - Base Study Placebo | Group 4 - Quadrivalent Human Papillomavirus Vaccine Extension
Serious Adverse Events (participants affected / at risk) | 50/2673 | 4/299 | 45/2672 | 5/801
Other Adverse Events (participants affected / at risk) | 2458/2673 | 276/299 | 2331/2672 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine (N=2673) | Group 2 - Base Study Monovalent HPV (Type 16) Vaccine (N=299) | Group 3 - Base Study Placebo (N=2672) | Group 4 - Quadrivalent Human Papillomavirus Vaccine Extension (N=801)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Allergy to vaccine (Immune system disorders) | 0 | 0 | 0 | 1
Anogenital warts (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0
Endometritis decidual (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 2 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 2 | 0 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Accidental poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 16 | 2 | 21 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Facial palsy (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 1 | 0
Cervix dystocia (Pregnancy, puerperium and perinatal conditions) | 4 | 0 | 0 | 0
Failed induction of labor (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Failed trial of labor (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Fetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Fetal malposition (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 3 | 0
Premature labor (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 1 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
Prolonged labor (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Base Study Quadrivalent Human Papillomavirus Vaccine (N=2673) | Group 2 - Base Study Monovalent HPV (Type 16) Vaccine (N=299) | Group 3 - Base Study Placebo (N=2672) | Group 4 - Quadrivalent Human Papillomavirus Vaccine Extension (N=0)
Abdominal pain (Gastrointestinal disorders) | 88 | 8 | 81 | 0
Abdominal pain upper (Gastrointestinal disorders) | 82 | 5 | 87 | 0
Diarrhea (Gastrointestinal disorders) | 105 | 9 | 96 | 0
Dyspepsia (Gastrointestinal disorders) | 17 | 5 | 16 | 0
Gastritis (Gastrointestinal disorders) | 22 | 4 | 13 | 0
Nausea (Gastrointestinal disorders) | 210 | 23 | 174 | 0
Toothache (Gastrointestinal disorders) | 48 | 4 | 40 | 0
Vomiting (Gastrointestinal disorders) | 62 | 9 | 56 | 0
Asthenia (General disorders) | 29 | 7 | 25 | 0
Fatigue (General disorders) | 73 | 12 | 102 | 0
Malaise (General disorders) | 47 | 3 | 40 | 0
Pain (General disorders) | 19 | 3 | 26 | 0
Pyrexia (General disorders) | 436 | 33 | 348 | 0
Gastroenteritis (Infections and infestations) | 17 | 3 | 18 | 0
Influenza (Infections and infestations) | 124 | 18 | 113 | 0
Nasopharyngitis (Infections and infestations) | 185 | 22 | 166 | 0
Pharyngitis (Infections and infestations) | 32 | 3 | 31 | 0
Sinusitis (Infections and infestations) | 22 | 3 | 18 | 0
Tonsillitis (Infections and infestations) | 26 | 2 | 29 | 0
Upper respiratory tract infection (Infections and infestations) | 36 | 9 | 42 | 0
Vulvovaginal candidiasis (Infections and infestations) | 10 | 4 | 16 | 0
Procedural pain (Injury, poisoning and procedural complications) | 4 | 3 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 0 | 25 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 68 | 10 | 63 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 14 | 3 | 12 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 49 | 6 | 54 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 55 | 7 | 57 | 0
Dizziness (Nervous system disorders) | 123 | 18 | 114 | 0
Headache (Nervous system disorders) | 802 | 103 | 76 | 0
Migraine (Nervous system disorders) | 23 | 3 | 15 | 0
Somnolence (Nervous system disorders) | 30 | 0 | 32 | 0
Insomnia (Psychiatric disorders) | 35 | 2 | 23 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 106 | 11 | 100 | 0
Pelvic Pain (Reproductive system and breast disorders) | 14 | 4 | 22 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 59 | 6 | 40 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 26 | 3 | 15 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 109 | 14 | 116 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 5 | 3 | 10 | 0
Injection site erythema (General disorders) | 659 | 84 | 450 | 0
Injection site haematoma (General disorders) | 94 | 6 | 97 | 0
Injection site hypersensitivity (General disorders) | 27 | 9 | 22 | 0
Injection site pain (General disorders) | 2281 | 242 | 2014 | 0
Injection site pruritus (General disorders) | 109 | 12 | 80 | 0
Injection site reaction (General disorders) | 22 | 4 | 17 | 0
Injection site swelling (General disorders) | 694 | 70 | 413 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.